CLINICAL TRIAL: NCT03755882
Title: Clinical Comparison of Two Marketed Reusable Cosmetic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6286
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2020-01-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Female subjects between the ages of 18 to 29 years who are habitual reusable soft cosmetic contact lens wearers will be randomized into one of two lens sequences.
  Interventions: Device: ACUVUE® DEFINE™ Vivid Style; Device: LACELLE™ Sparkling Brown
- CONTROL/TEST (Experimental): Female subjects between the ages of 18 to 29 years who are habitual reusable soft cosmetic contact lens wearers will be randomized into one of two lens sequences.
  Interventions: Device: ACUVUE® DEFINE™ Vivid Style; Device: LACELLE™ Sparkling Brown

INTERVENTIONS:
Device: ACUVUE® DEFINE™ Vivid Style — TEST Lens
  Other Names: etafilcon A
Device: LACELLE™ Sparkling Brown — CONTROL Lens
  Other Names: helifilcon A

SUMMARY:
This will be a 4-visit, multi-site, randomized, brand-masked, bilateral, 2×2 crossover study. If a subject is found to meet all eligibility criteria, they will be randomized to one of two lens wear sequences. Each lens type will be worn for approximately 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol (ie, willing to wear only the study lenses and not use habitual lenses during the study).
  3. Females between 18 and 29 (inclusive) years of age at the time of screening
  4. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -2.00 D to -7.00 D (inclusive) in each eye.
  5. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye.
  6. Have spherical best corrected logMAR visual acuity (VA) of 0.18 or better in each eye.
  7. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report.
  8. Must be habitual reusable (2 week, or monthly), cosmetic contact lenses wearers.
  9. The subject must be willing to be photographed and/or video-taped

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating
  2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion).
  3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion).
  4. Any previous, or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.)
  5. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment.
  6. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician).
  7. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion).
  8. Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Zhongshan Ophthalmic Center, Guanzhou, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 subjects were enrolled into this study. Of those enrolled 45 were dispensed at least 1 study lens. Of those dispensed, 41 subjects completed the study while 4 were discontinued.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 23 | 22
Completed | 19 | 22
Not Completed | 4 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Unsatisfactory Lens Fitting Test Article | 3 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 19 | 22
Completed | 19 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: All subjects dispensed a study lens
Arm/Group | Total
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.6 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 45
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 45

OUTCOME MEASURES:

1. Primary Outcome: Visual Performance
Description: Monocular visual performance (logMAR) was evaluated under 3 conditions (1.high luminance and high contrast, 2. High Lumiance Low Contrast and 3. Low Luminance High Contrast with distance goggles) at 4 meters using Early Treatment Diabetic Retinopathy Study (ETDRS) charts. Letter-by-letter results were calculated to ascertain the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: Up to 2-Week Follow-up
Population: All subjects who had successfully completed all visits.
Measure: Mean (Standard Deviation); unit: logMAR Units
Units Other Than Participants: Eyes
Groups:
- Test (Etafilcon A): Subjects that wore the Test lens in either the first or second period of the study.
- Control (Hefilcon A): Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test (Etafilcon A) | Control (Hefilcon A)
Number analyzed (Participants) | 45 | 41
Number analyzed (Eyes) | 90 | 82
logMAR Units
  High Luminnance Low Contrast: number analyzed (Participants) | 43 | 41
  High Luminnance Low Contrast | 0.40 (0.074) | 0.38 (0.086)
  High Luminance High Contrast | -0.09 (0.053) | -0.10 (0.059)
  Low Luminance High Contrast with Distance Goggles | -0.10 (0.055) | -0.09 (0.055)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 5 weeks per subject.
Arm/Group | Test (Etafilcon A) | Control (Hefilcon A)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT03755882/Prot_SAP_000.pdf